CLINICAL TRIAL: NCT05290285
Title: Efficacy and Tolerability of a Specific Blend of Amino Acids in Patients With Anorexia Nervosa Treated in a Hospital Setting. Double-blind Randomized Study Versus Placebo
Brief Title: Amino Acids in Patients With Anorexia Nervosa: Double-blind Randomized Study Versus Placebo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Villa Garda Hospital (Other)
Collaborators: University of Milan (Other); Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Riccardo Dalle Grave, M.D., Villa Garda Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ATAN/22
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa
Keywords: lean body mass; amino-acids
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: A 13-week randomized double-blind placebo-controlled study.
  Patients will be randomized to EAA supplementation or placebo supplementation upon admission. Randomisation will be carried out by an independent external figure adopting the following stratification:
  Group 1: BMI <= 15.2 & age <= 20 Group 2: BMI > 15.2 & age <= 20 Group 3: BMI <= 15.2 & age > 20 Group 4: BMI > 15.2 & age > 20
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EAA supplementation (Experimental): The EAA blend consists of a complex blend of essential amino acids, including some precursors of neurotransmitters that are important for regulating mood. In particular, phenylalanine, a precursor of tyrosine (non-essential amino acid) is involved in the biosynthesis of catecholamines (noradrenaline, adrenaline, dopamine) and tryptophan is the precursor of serotonin. Furthermore, the amino acids present in the mixture and the precursors of the Krebs cycle (citrate, malate, succinate) are able to stimulate mitochondrial bioenergetics by improving metabolism and muscle function.
  The EAA blend will be administered orally at 4.5 g twice daily (two sachets of Amino-Ther Pro per day).
  Interventions: Dietary Supplement: Amino-Ther Pro
- Placebo (Placebo Comparator): Placebo is an isocaloric product containing maltodextrins instead of amino acids (Acquilani et al., 2011). The placebo will be administered orally 4.5 g twice daily.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Amino-Ther Pro — Food supplements
  Arms: EAA supplementation
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
Amino acids (AAs) are crucial for protein synthesis, in influencing nutritional status, as sources of vital elements (e.g., nucleotides, neurotransmitters) and as signal molecules for the modulation of gene expression and epigenetic mechanisms. Data on the role of amino acids in underweight patients with anorexia nervosa (AN) are unknown. This study aims to evaluate whether a blend of essential amino acids (EAA) could influence the change in lean body mass (LBM) in patients with AN during weight restoration, treated with intensive inpatient enhanced cognitive behavior therapy (CBT-E). A total of 92 patients will be randomized to EAA supplementation or placebo supplementation upon admission to inpatient treatment. LBM, but also body weight, specific and general psychopathology, impairment assessment will be assessed at baseline and after 13 weeks of treatment.

DETAILED DESCRIPTION:
Nutrition is one of the main determinants of health. Among the three primary macronutrients, proteins - specifically, their quantity and quality (i.e., their specific amino acid profile) - play a crucial role in regulating metabolic health and longevity. Amino acids (AAs) are crucial not only for protein synthesis and influencing nutritional status but also as sources of vital elements (e.g., nucleotides, neurotransmitters) and as signal molecules for the modulation of gene expression and epigenetic mechanisms. To our knowledge, only one study was conducted on underweight patients with anorexia nervosa (AN). The study design was to compare the efficacy of the semi-essential amino acid L-tyrosine (100 mg/kg/day) versus a placebo supplement. Tyrosine reduced reaction time and test duration in memory tasks and improved mood. However, to date, no studies have evaluated the effect of supplementation with amino acids in patients with anorexia nervosa who undergo specialist treatment aimed at weight recovery and remission from psychopathology.

The study has the primary aim of evaluating the effectiveness of supplementation with essential amino acids (EAA) on the change in lean body mass (LBM) with weight recovery in patients with AN treated with specialist treatment for eating disorders, compared to placebo supplementation. The secondary aims of the study are to evaluate the effectiveness of EAA supplementation on physical fitness, weight recovery, change of the general and eating disorder psychopathology, and psychosocial impairment, compared to placebo supplementation.

A 13-week randomized double-blind placebo-controlled study design will be used.

Patients will be randomized to EAA supplementation or placebo supplementation upon admission. Randomization will be carried out by an independent external figure adopting the following stratification:

Group 1: Body Mass Index (BMI) <= 15.2 & age <= 20 Group 2: BMI > 15.2 & age <= 20 Group 3: BMI <= 15.2 & age > 20 Group 4: BMI > 15.2 & age > 20 Treatment will involve a 13-week inpatient or a 13-week day hospital. Follow-up will be performed for both groups at 24 weeks. Considering that it will not be possible to carry out a closed follow-up, we will give the possibility to those who have taken the mixture of EAA to continue this treatment after the end of inpatient or day-hospital, for other 24 weeks, to evaluate the potential long-term maintenance of the treatment.

The study is performed at the Nutritional Rehabilitation Unit of the Villa Garda Hospital - Italy.

The supervision of the diagnostic evaluation and treatment is carried out weekly by the Director of the Nutritional Rehabilitation Unit of the Villa Garda Hospital.

Study participants will be recruited from patients who meet the diagnostic criteria for AN, assessed with the Eating Disorder Examination (EDE.17) interview, consecutively admitted at the Nutritional Rehabilitation Unit of the Villa Garda Hospital. All participants will meet the appropriateness criteria of hospitalization established by the Veneto Region and described in table 1 of Annex B of DGR 94/2012.

On the entry day into the Nutritional Rehabilitation Unit, the patient will meet a unit physician for the medical history collection, the physical examination, and the prescription of humoral and instrumental examinations. On this occasion, the enrollment phase will take place which will include the complete collection of data for the compilation of the Data Collection Form. At the end of the data collection, if the criteria for inclusion in the study are met, the patient will receive detailed information on:

* Procedures and objectives of the study
* Purposes, methods, inconveniences, risks, and benefits that the study may entail
* Freedom to participate and withdraw from the study without affecting subsequent treatment
* Compensation procedures and treatment of any damages deriving from participation in the study.

Before requesting to sign the informed consent and the possibility of using (and having consent to use) the information collected during the trial, the patient will be given a statement to read containing detailed information on the study.

If the patient, or in the case of a minor patient, his/her parents (s), and/or legal guardians (s), agrees to participate in the study, he/she will sign the informed consent form and the authorization to process personal and sensitive data.

If the patient meets the criteria for inclusion in the study but refuses to participate in the study, he/she will continue the intensive rehabilitation treatment applied at the Nutritional Rehabilitation Unit of the Villa Garda Hospital.

After the interview and signing the informed consent and data processing, the patient will be randomized to EAA supplementation or placebo supplementation. Both arms will receive enhanced cognitive behavior therapy (CBT-E).

The intensive CBT-E applied at the Nutritional Rehabilitation Unit of the Villa Garda Hospital has been described in national and international publications. The treatment is based on the transdiagnostic cognitive-behavioral theory and therapy of eating disorders developed by the Center for Research on Eating Disorders and Obesity of the University of Oxford.

The inpatient treatment includes 13 weeks, followed by seven weeks of day-hospital, and is divided into four phases that are individualized to address the maintenance mechanisms of the eating disorder psychopathology operating in the individual patient.

* Phase One - Starting Well. This phase aims to engage the patient, educate him about his eating disorder, build the Personalized Formulation, start the collaborative weight measurement and use the Monitoring Records and the Eating Problem Check List (EPCL) questionnaire. During this phase, the patient is encouraged to make maximum behavioral change, including starting the weight regain process, if indicated.
* Phase Two. In this phase, a formal assessment of the progress and obstacles to change and of the possible presence of external maintenance mechanisms is performed to plan the next phase of treatment.
* Phase Three. The precise content of this phase is dictated by the specific psychopathology operating in the patient and the treatment becomes very individualized. In typical cases, negative body image, calorie and cognitive dietary restriction, events and emotions affecting nutrition, and, in a subset of patients, one or more of the external maintenance mechanisms identified in Phase Two are addressed in specific modules of the extended version of the treatment. At this stage, the underweight patient in most cases reaches his BMI goal and starts practicing weight maintenance. Towards the end of this phase, backward steps and mental states are also addressed to learn to decentralize oneself from the mental state of the eating disorder, to prevent relapse.
* Phase Four - Ending Well. This phase aims to conclude the treatment well and prepare the transition to outpatient therapy. For this purpose, a written maintenance plan is created, in collaboration with the patient, in which the residual problems are to be faced and the procedures to continue to be used, the strategies and methods to prevent relapse, the ways of organizing life after discharge and post-admission therapy.

The nutritional rehabilitation protocol of the Villa Garda Hospital applied to underweight patients with AN is as follows:

* The weight goal to be achieved is a BMI ≥ 19.
* The expected speed of weight recovery is between 1 and 1.5 kg per week.
* The daily calorie content of the meal plan is established collaboratively with the patient in the first as follows:

  * Week 1: Menu A (1,500 kcal)
  * Week 2: Menu B (2,000 kcal)

Afterward:

* If the weight increases between 1 and 1.5 kg per week the meal plan is maintained with the same calorie content as the previous week.
* If the weight increases by less than 1 kg per week, the kcal of the food plan is increased by 500 kcal per day. For example, from Menu B to Menu C (2500 kcal) or from Menu C to Menu D (3000 kcal)
* If the weight increases by more than 1.5 kg per week, the kcal of the food plan must be reduced by 250 kcal per day. For example, from Menu C to Menu B / C (2250 kcal)
* When the patient reaches a BMI of 19, the goal of the program is to identify a weight range of 3 kg that it can be without adopting a calorie dietary restriction. In most patients, weight maintenance occurs with a diet between 2000 (Menu B) and 2500 kcal (Menu C).

  * Physical activity proposed in the rehabilitation program All patients above the BMI of 15 do two 30-minute sessions per week of calisthenics followed by a physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of anorexia nervosa
* Age between 16 and 50 years
* Written informed consent

Exclusion Criteria:

* Schizophrenia or other psychotic disorders
* Diagnosis of bulimia nervosa
* Current and ongoing substance use disorder
* Medical complications capable of hindering the interpretation of the results (e.g. a a medical disease that induces weight loss)
* Presence of physical treatments (including drugs) hindering the interpretation of the results (e.g. chemotherapy for cancer)
* Being pregnant or intending to become pregnant during treatment

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Lean body mass | From baseline (admission to inpatient) to end of hospitalization (after 13 weeks)
  Percentage change in patient's lean body mass with weight gain at the end of hospital treatment, measured using the DXA (Prodigy Primo Lunar, A223040501, General Electric Company, Madison. WI 53707-7550, USA-EnCORE TM 2009 (v13.31) software)

SECONDARY OUTCOMES:
Physical fitness | From baseline (admission to inpatient) to end of hospitalization (after 13 weeks)
  Change in physical fitness measured using the Eurofit Physical Fitness Test Battery (EPFTB) (EUROFIT Strasbourg: Council of Europe; 1993
Body weight | From baseline (admission to inpatient) to end of hospitalization (after 13 weeks)
  Change in body weight measured using the Seca Digital Wheelchair Scale Model 664 [Seca, Hamburg, Germany]
Eating disorder psychopathology | From baseline (admission to inpatient) to end of hospitalization (after 13 weeks)
  Change in eating disorder psychopathology measured using the Eating Disorder Examination Questionnaire (EDE-Q) (Calugi, Milanese, et al., 2017; Fairburn & Beglin, 2008).
General psychopathology | From baseline (admission to inpatient) to end of hospitalization (after 13 weeks)
  Change in general psychopathology measured using the Brief Symptom Inventory (BSI) (De Leo, Frisoni, Rozzini, & Trabucchi, 1993; Derogatis & Spencer, 1982).
Clinical impairment | From baseline (admission to inpatient) to end of hospitalization (after 13 weeks)
  Change in clinical impairment measured using the Clinical Impairment Assessment (CIA) (Bohn et al., 2008; Calugi et al., 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Dalle Grave, MD, Principal Investigator — Villa Garda Hospital
Locations (1):
- Department of Eating and Weight Disorders, Villa Garda Hospital, Garda, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not available for privacy reasons

REFERENCES:
- [Background] Dalle Grave R, Calugi S, Conti M, Doll H, Fairburn CG. Inpatient cognitive behaviour therapy for anorexia nervosa: a randomized controlled trial. Psychother Psychosom. 2013;82(6):390-8. doi: 10.1159/000350058. Epub 2013 Sep 20. PMID 24060628
- [Background] El Ghoch M, Pourhassan M, Milanese C, Muller MJ, Calugi S, Bazzani PV, Dalle Grave R. Changes in lean and skeletal muscle body mass in adult females with anorexia nervosa before and after weight restoration. Clin Nutr. 2017 Feb;36(1):170-178. doi: 10.1016/j.clnu.2015.10.006. Epub 2015 Oct 28. PMID 26560758
- [Background] Buondonno I, Sassi F, Carignano G, Dutto F, Ferreri C, Pili FG, Massaia M, Nisoli E, Ruocco C, Porrino P, Ravetta C, Riganti C, Isaia GC, D'Amelio P. From mitochondria to healthy aging: The role of branched-chain amino acids treatment: MATeR a randomized study. Clin Nutr. 2020 Jul;39(7):2080-2091. doi: 10.1016/j.clnu.2019.10.013. Epub 2019 Oct 18. PMID 31672329
- [Background] Israely M, Ram A, Brandeis R, Alter Z, Avraham Y, Berry EM. A Double Blind, Randomized Cross-Over Trial of Tyrosine Treatment on Cognitive Function and Psychological Parameters in Severe Hospitalized Anorexia Nervosa Patients. Isr J Psychiatry. 2017;54(3):52-58. PMID 29735813
- [Background] Fairburn CG, Cooper Z, Shafran R. Cognitive behaviour therapy for eating disorders: a "transdiagnostic" theory and treatment. Behav Res Ther. 2003 May;41(5):509-28. doi: 10.1016/s0005-7967(02)00088-8. PMID 12711261
- [Derived] Dalle Grave R, Calugi S, Ruocco C, Chimini M, Segala A, Ragni M, Carruba M, Valerio A, Nisoli E. Efficacy and tolerability of a specific blend of amino acids in patients with anorexia nervosa treated in a hospital setting: study protocol for a randomized controlled trial. Trials. 2023 Feb 9;24(1):104. doi: 10.1186/s13063-023-07120-7. PMID 36759873